CLINICAL TRIAL: NCT06980753
Title: Continuous Steroid Monitoring in Interstitial Fluid With Wearable and Nanoparticle-enhanced Biosensors for Improved Management of Adrenal Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Swiss Federal Institute of Technology in Zurich (ETH Zurich) (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Madson Queiroz de Almeida, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Adrenal biossensor 01
Record Dates: First submitted 2025-04-25; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Cushing Syndrome; Primary Aldosteronism; Adrenal Insufficiency
Keywords: Aldosterone; Cortisol; Biossensor; Interstitial fluid; Adrenal insuficiency; Cushing syndrome
MeSH Terms: conditions — Cushing Syndrome; Hyperaldosteronism; Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interstitial fluid collection and biossensor use (Experimental)
  Interventions: Device: Participants will use the biossensor for 48 h

INTERVENTIONS:
Device: Participants will use the biossensor for 48 h — Participants will use the biossensor for 48 h

SUMMARY:
The goal of this project is to provide novel technology that will pave the way from the present single-point (analogue) endocrinology towards continuous cortisol and aldosterone monitoring with full time resolution. Current endocrine practice relies on occasional and often random determination of hormone level or functional tests that require a clinical setting. These measurements include sample extraction and analysis in a clinical laboratory rendering such tests laborious and expensive. Most importantly, through the individual variations of hormone oscillation and spatiotemporal distribution of hormones, infrequent hormone measurements have limited diagnostic and prognostic value as the dynamic changes are not captured and relevant intra-individual variability occurs. A requirement for this vision are sensing solutions capable to track hormone dynamics over prolonged periods at high patient comfort (e.g., at home), as targeted by this research proposal. This project has the overarching goals of (1) establishing dynamic interstitial aldosterone and cortisol monitoring as reliable diagnostic tool for cortisol and aldosterone excess or deficiency, and (2) develop a wearable molecular sensing device to detect them accurately.

DETAILED DESCRIPTION:
To trace steroid dynamics in a routine setting, the choice of body fluid is critical, as it dictates the ease and frequency of collection that is tolerated by individuals. While the gold standard is based on blood assay, several body fluids can be accessed minimally invasive, including urine, sweat, breath, saliva and interstitial fluid. More promising for steroid monitoring is interstitial fluid, as it closely mirrors the composition of blood plasma due to continuous mass transfer. In fact, this has been demonstrated just last year using a subcutaneously implanted micro-dialysis catheter that collected interstitial fluid with an infusion pump. Worn around the waist, samples were collected for 24 hours in 214 volunteers and analysed offline by liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS). That way, cortisol was accurately traced and followed a similar dynamic in tissue (i.e., interstitial fluid) compared to blood plasma. On this basis, disease-related differences were detected, for example, elevated cortisol concentrations in a patient suffering from Cushing syndrome. Yet, extended investigations of the aldosterone and cortisol dynamics in interstitial fluid under different clinical scenarios of hormone excess and deficiency, and validation against serum measurements are required to establish this method for diagnostic and treatment purposes.

This project has the overarching goals of (1) establishing dynamic interstitial aldosterone and cortisol monitoring as reliable diagnostic tool for cortisol and aldosterone excess or deficiency, and (2) develop a wearable molecular sensing device to detect them accurately. In the work package 1 (Characterization of interstitial cortisol and aldosterone concentrations): The diagnostic utility of cortisol and aldosterone measurement in the interstitial fluid will be assessed by comparative quantification to serum concentration by LC-MS/MS. Therefore, interstitial fluid and blood will be collected in healthy individuals and patients during the morning (when cortisol and aldosterone reach the highest levels) and during dynamic tests to investigate adrenal diseases, such as ACTH (cosyntropin) stimulation test (which evaluates the peak cortisol response following an exogenous stimulus) and saline infusion test (which evaluates aldosterone suppression following volume and sodium overload). Since continuous interstitial fluid is not yet possible, commercially available hollow microneedle devices will be used for single timepoint extraction.

Main hypothesis 1: Cortisol and aldosterone concentrations in interstitial fluid reflect sufficiently well blood serum concentrations to reliably indicate normal steroid secretion and the onset of cortisol and aldosterone disorders.

In this first step, the investigators will perform a pairwise comparison of cortisol and aldosterone concentrations in interstitial fluid with serum measurements. This study will be submitted to the responsible Ethics Committees of USP. The written informed consent will be signed by all participants. The investigators will evaluate 150 individuals, including healthy controls and patients with adrenal hyper- and hypofunction referred for evaluation in the outpatient clinic of the Adrenal Unit, Division of Endocrinology, USP. Clinical and hormone evaluation of the enrolled patients with adrenal disorders will follow the standard guidelines of the Endocrine and European Society of Endocrinology. All healthy controls (without a previous diagnosis of adrenal disease) will have an appointment to fill out a questionnaire of medical history and to collect blood tests.

Individuals (males and females) older than 18 years will be eligible for inclusion. Patients covering a broad spectrum of adrenal diseases will be recruited: cortisol and aldosterone deficiency (primary adrenal insufficiency), cortisol excess (Cushing syndrome) and aldosterone excess (primary aldosteronism). A single timepoint of each participant will be evaluated in the morning following overnight fasting and without morning medication. This baseline evaluation will allow to sample material with normal, low (adrenal insufficiency) and high (Cushing's syndrome and primary aldosteronism, respectively) adrenal steroid content. In addition, ACTH (intravenous 250 µg cosyntropin) stimulation test will be performed in healthy controls and patients under investigation of adrenal insufficiency and primary aldosteronism to correlate interstitial aldosterone and cortisol levels with the peak of serum cortisol and aldosterone after 1h of ACTH stimulus. The saline infusion test (intravenous 2 liter of 0.9% saline over 4h) will be performed in the patients under investigation for primary aldosteronism. These dynamic tests will be performed in a dynamic test room in the outpatient clinic, which counts with a team of endocrinologist, nurse, and technicians trainned for endocrine dynamic evaluation. Exclusion criteria will be as follows: use of estrogen-containing oral contraceptive medication within the past 6 weeks; pregnancy or lactation; use of oral, inhaled, parenteral, or topical glucocorticoids within the past 30 days. Basal sample collection and dynamic tests will be performed at fasting between 8 am to 10 am.

In work package 2 (Establish hollow microneedles for continuous interstitial fluid extraction) the investigators will demonstrate the direct printing of polymer-based microneedles with optimized mechanical and fluid dynamic properties onto microfluidic chips for continuous interstitial fluid extraction: A wearable patch for continuous interstitial fluid extraction will be developed. It will consist of hollow microneedles directly 3D-printed onto microfluidic chips. The needles will be based on biocompatible polymer to minimize skin irritation during prolonged application, while the microfluidic chips will be fabricated by scalable micromachining. Needle penetration depth and stability will be tested on human skin analogues, while fluid dynamic properties and extraction rates are assessed with artificial interstitial fluid.

Main hypothesis 2: Interstitial fluid can be accessed non-invasively and continuously over extended periods with hollow microneedles based on biocompatible materials.

In work package 3 (Establish and utilize steroid biosensor based on aptamer-functionalized nanoparticles Biosensors for real-time and continuous quantification of cortisol and aldosterone in interstitial fluid will be developed) the investigators will investigate aptamer-functionalized nanoparticles decorated with plasmonic clusters to bind steroids followed by their release through light stimulation to yield selective and rapidly reversible sensing for continuous biomarker monitoring: The receptor will be based on aptamers that are immobilized on nanoparticles to detect analyte binding and quantify concentrations electrochemically. The nanoparticles will be populated also with plasmonic clusters (e.g., Au or Ag) to serve as heat-source when activated by light to trigger analyte release. The cluster-loaded nanoparticles will be designed at controlled composition and size by flame-aerosol technology, and deposited directly onto microfluidic platforms as porous films.

Main hypothesis 3: Aptamers will enable a selective binding of cortisol and aldosterone. By immobilizing these aptamers on nanoparticles, binding events are recognized during electrochemical sensing. The recovery of the sensor will be enabled by exploiting thermoplasmonic effects when exposed to light, to trigger the release of the analyte by local heating. The porous film morphology of the sensing film enables rapid mass transfer of the analyte.

Based on the performance requirements identified by USP under WP1, biosensor will be developed at ETH Zurich to perform real-time and continuous quantification of cortisol and aldosterone to provide longitudinal profiles.

In work package 4 (Clinical validation of wearable aldosterone and cortisol sensor in adrenal disease) the wearable biosensor developed under WP2 and WP3 will be evaluated as a diagnostic tool for adrenal disease. The written informed consent will be signed by all participants after study approval by the Ethics Committees of USP. All participants will be evaluated in the outpatient clinic of the Adrenal Unit, Division of Endocrinology, USP. The dynamic tests (ACTH stimulation and saline infusion tests) will be performed in a dynamic test room in the outpatient clinic, which counts with a team of endocrinologist, nurse, and technicians trainned for endocrine dynamic evaluation. Clinical and hormone evaluation of the enrolled patients with adrenal disorders will follow the standard guidelines of the Endocrine and European Society of Endocrinology. All healthy controls (without a previous diagnosis of adrenal disease) will have an appointment to fill out a questionnaire of medical history and to collect blood tests. Participants will be asked to maintain a regular bedtime, abstain from alcohol, and to avoid any strenuous physical activity before and during biosensor use. Moreover, participants will be asked to complete an activity diary, including records of food type and timing, sleep timing, and any unexpected event during the time wearing the biosensor. 96 prototypes will be transferred from ETH to USP and tested during 48h in the following subgroups under the specified conditions:

Controls: 32 healthy volunteers will be tested during ACTH (intravenous 250 µg cosyntropin) stimulation test at the morning of the second day of continuous cortisol and aldosterone measurements.

Cortisol disorders: 32 patients with adrenal insufficiency or Cushing syndrome will be tested during a ACTH stimulation test on the second day of continuous steroid measurements.

Primary aldosteronism: 32 patients under investigation for primary aldosteronism will be continuously monitored. The saline infusion test (intravenous 2 L 0.9% saline over 4h) will be performed in the second day of continuous measurements of aldosterone and cortisol.

As a further step of biosensor validation , blood samples will be collected at the morning (8 am to 10 am) and during the dynamic tests (ACTH stimulation and saline infusion tests) to measure cortisol and aldosterone by LC-MS/MS. Correlation between serum cortisol and aldosterone concentrations and the interstitial measurements obtained with the biosensor will be analyzed. During the time of biosensor use, the total area under the curve (AUC), the morning peak and the night nadir of cortisol and aldosterone interstitial measurements will be calculated for each patient. These measures will be compared between patients with adrenal disease and healthy controls to determine the diagnostic applications of interstitial cortisol and aldosterone dynamics.

These four challenges will be approached by an interdisciplinary team at USP (clinical) and ETH (engineering) through four work packages (WP) focusing on interstitial fluid characterization (WP1), microneedle sampler (WP2), biosensing (WP3) and clinical validation (WP4) of the resulting wearable prototype.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (males and females) older than 18 years;
* Patients with primary adrenal insuffiency (cortisol and aldosterone deficiency);
* Patients with Cushing Syndrome (cortisol excess)
* Patients with Primary Aldosteronism (aldosterone excess)

Exclusion Criteria:

* Use of estrogen-containing oral contraceptive medication within the past 6 weeks;
* Pregnancy or lactation;
* Use of oral, inhaled, parenteral, or topical glucocorticoids within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The total area under the curve (AUC) of aldosterone and cortisol levels measured over 48 hours using the biossensor | 8 weeks
  It is important to note that the units of concentration for aldosterone (ng/dl) and cortisol (mcg/dl) do not influence the calculation of the AUC

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo - General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No